CLINICAL TRIAL: NCT06440278
Title: Multisite Feasibility of BA-HD: An Integrated Depression and Behavioral Risk Factor Reduction Coaching Program Following Acute Coronary Syndrome
Brief Title: Healthy Heart Habits-2
Acronym: HHH-2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Principal Investigator, Emily C. Gathright, PhD, Research Scientist, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34HL165716-01A1 (NIH)
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Activation for Health and Depression (Experimental)
  Interventions: Behavioral: Behavioral Activation for Health and Depression (BA-HD)
- Enhanced Usual Care (Active Comparator)
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Behavioral Activation for Health and Depression (BA-HD) — BA-HD includes 8 - 10 sessions delivered over 10-12 weeks. Sessions use behavioral activation techniques to connect patient core values with goal-setting targeting activities that improve mood, alongside personalized adjustments to cardiovascular health behaviors (i.e., tobacco cessation, medication adherence, physical activity, diet, and sleep). Educational materials and commercially available tools like activity trackers, pillboxes, and portion control aids will accompany the goal-setting process to facilitate behavior change.
  Arms: Behavioral Activation for Health and Depression
Other: Enhanced Usual Care — Patients will receive depression and heart disease education, as well as a list of local mental health resources.
  Arms: Enhanced Usual Care

SUMMARY:
Sixty adults who have experienced acute coronary syndrome within the past 2-12 months from three states (Rhode Island, North Carolina, Minnesota) will be randomized to either (1) a coaching program for depressed mood and health behavior change (Behavioral Activation for Health and Depression; BA-HD), or (2) Enhanced Usual Care. This study will evaluate the feasibility and acceptability of study procedures and BA-HD, and establish protocol and measurement harmonization across three sites in preparation for a future multi-site efficacy trial.

DETAILED DESCRIPTION:
Acute coronary syndrome (ACS) represents a significant public health burden, with the most recent estimates suggesting that over 1 million U.S. adults experience ACS per year. As individuals are acutely surviving ACS more often, the associated disease burden is increasing for both the healthcare system and the individual living post-ACS.

Poor engagement in health behaviors post-ACS contributes to risk for recurrent ACS and mortality. Modifiable behavioral contributors include smoking, medication non-adherence, physical inactivity, and poor diet. Approximately 20% of post-ACS adults experience depression and depression is associated with worse engagement in critical health behaviors, which in turn, increases subsequent progression of cardiovascular disease. Treatment of depression alone improves, but does not eliminate, behavioral nonadherence. Behavioral Activation is a robust counseling treatment for depression with evidence of improvements in depressive symptoms across varied populations (including those with medication conditions). BA seeks to improve mood by increasing environmental reinforcement through collaborative, values-guided setting of "activation goals." The goal setting focus and structure of BA allows for seamless integration of health behavior targets and thus offers a potential framework to integrate depression and health behavior treatment. BA-HD may be a useful strategy to depression and multiple health behavior improvement post-ACS. However, this possibility requires further testing.

The purpose of this study is to examine the feasibility and acceptability of a multisite pilot randomized controlled trial and test the initial potential effects of the intervention (BA-HD) on cardiovascular health and depressive symptoms relative to an Enhanced Usual Care control condition. Participants will be randomly assigned to either 12 weeks of tele-delivered BA-HD) or Enhanced Usual Care (i.e., one session of depression and heart disease education and provision of community mental health resources).

Primary endpoints are feasibility of multisite recruitment procedures (e.g., recruitment rates at each site), feasibility of intervention and control procedures (e.g., percent of enrolled participants who complete the study), study retention (e.g., percent of participants who complete 3 month follow-up), and acceptability of intervention content and intervention delivery and control procedures. The investigators hypothesize that the intervention content and delivery will be 1) feasible and 2) acceptable. The investigators will also examine changes in cardiovascular health, depressive symptoms, medication adherence, affect, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Medical chart-documented ACS (diagnosis of unstable angina, ST or non-ST elevation myocardial infarction) occurrence within the past 2-12 months.
* Post-ACS depressed mood defined as a Patient Health Questionnaire(PHQ)--9 score ≥ 10 upon screening,
* Non-adherence to and willingness to implement changes to ≥1 health behavior based on screening of:

  1. Smoking/Tobacco exposure,
  2. Physical Activity,
  3. Diet,
  4. Sleep health,
  5. Medication adherence
* English-language fluency
* Resides within 90 minutes (driving time) of each site with no plans to relocate beyond that range during study participation
* Access to a telephone and/or videoconferencing capability
* Has primary care provider
* Address at which packages can be received

Exclusion Criteria:

* Chart indication of significant cognitive impairment (e.g., chart-documented dementia), Current exacerbation of serious mental illness,
* Suicidality,
* Hearing impairment that prevents telephone/video communication for intervention and assessment purposes,
* Current hospice care, and
* Current engagement in cardiac rehabilitation or other regular counseling treatment targeting depression or health behavior change

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Recruitment feasibility | Baseline
  Number of participants randomized per month of recruitment
Study retention | Week 26
  Proportion of randomized participants who complete the 6 month assessment.
Treatment engagement | Week 13
  Dose of treatment received (i.e., session attendance)
Treatment Acceptability | Week 13
  Client Satisfaction Questionnaire-8; Scores range from 8-32 with higher scores indicating greater treatment satisfaction.

SECONDARY OUTCOMES:
Cardiovascular Health | Week 13, Week 26
  Life's Essential 8 (LE8) Score; The LE8 classifies cardiovascular (CV) health across eight CV risk metrics: diet, physical activity, nicotine exposure, sleep health, weight, blood pressure, total cholesterol, and hemoglobin A1C. Each individual LE8 component is assigned a value ranging from 0 to 100. A total score is created by averaging each component score. Higher total scores reflect better overall CV health.
Depressive symptoms | Week 13, Week 26
  Patient Health Questionnaire-9; Scores range from 0 to 27; higher scores indicate greater depressive symptoms.
7 Day Moderate to Vigorous Physical Activity | Week 13, Week 26
  Minutes spent in moderate to vigorous physical activity from 7 day Actigraph wear
Self-Reported Moderate to Vigorous Physical Activity | Week 13, Week 26
  Minutes spent in moderate to vigorous physical activity over 7 days based on report from a 7 Day Physical Activity Recall interview
Self-Reported Diet | Week 13, Week 26
  Mediterranean Eating Pattern for Americans Questionnaire; Scores range from 0-16 with higher scores indicating greater consistency with mediterranean style diet
7-day point prevalence abstinence from smoking | Week 13, Week 26
  Self-report of no smoking, not even a puff, for 7 days; then Bio-chemically confirmed by carbon monoxide in a breath sample
Sleep duration | Week 13, Week 26
  Average hours of sleep per night over 7 nights assessed via 7 day Actigraph wear
Self-reported sleep duration | Week 13, Week 26
  Self-reported hours of sleep per night from the Pittsburgh Sleep Quality Index
Body Mass Index | Week 13, Week 26
  Body weight (kilograms)/ Height (meters squared)
Blood pressure | Week 13, Week 26
  Systolic and diastolic blood pressures (mmHg)
Non-HDL cholesterol | Week 13, Week 26
  mg/dL; measured via point of care testing
Hemoglobin A1C | Week 13, Week 26
  %; measured via point of care testing
Medication adherence (cholesterol regimen) | Week 13, Week 26
  DOSE-Nonadherence Extent of Nonadherence items will be used to assess self-reported medication adherence to cholesterol medication; scores range from 1-5.
Medication adherence (blood pressure regimen) | Week 13, Week 26
  DOSE-Nonadherence Extent of Nonadherence items will be used to assess self-reported medication adherence to blood pressure medication; scores range from 1-5
Medication adherence (blood glucose regimen) | Week 13, Week 26
  DOSE-Nonadherence Extent of Nonadherence items will be used to assess self-reported medication adherence to both oral and injectable medication (assessed separately) to manage blood glucose; scores range from 1-5
Major Adverse Cardiac Events | Week 26
  Composite of hospitalization for unstable angina, urgent coronary revascularization, and non-fatal myocardial infarction determined via participant inquiry and confirmed through electronic medical record review
All-cause mortality | Week 26
  Electronic medical record review
Health Behavior Engagement Composite | Week 13, Week 26
  A health behavior engagement composite score will be created that follows the LE8 scoring structure. LE8 component scores will be summed for physical activity, diet, combustible tobacco exposure, and sleep. Medication adherence will also be assigned a score ranging from 0 to 100 based on scaled DOSE-Nonadherence scores.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Gathright, PhD, Principal Investigator — The Miriam Hospital; Andrew Busch, PhD, Principal Investigator — Hennepin Healthcare Research Institute
Locations (3):
- United States (3):
  - Hennepin Healthcare Research Institute, Minneapolis, Minnesota
  - ECU Health, Greenville, North Carolina
  - The Miriam Hospital, Providence, Rhode Island